CLINICAL TRIAL: NCT04287036
Title: Objective Vision Evaluation of Two Cosmetic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6396
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible Subjects aged 18 to 39 years (inclusive) who are habitual soft contact lens wearers will be randomized into sequence, Test/Control
  Interventions: Device: JJVC Investigational Contact Lens; Device: 1-DAY ACUVUE® DEFINE® Radiant Sweet™
- Control/Test (Experimental): Eligible Subjects aged 18 to 39 years (inclusive) who are habitual soft contact lens wearers will be randomized into sequence, Control/Test.
  Interventions: Device: JJVC Investigational Contact Lens; Device: 1-DAY ACUVUE® DEFINE® Radiant Sweet™

INTERVENTIONS:
Device: JJVC Investigational Contact Lens — TEST
Device: 1-DAY ACUVUE® DEFINE® Radiant Sweet™ — CONTROL

SUMMARY:
This is a single visit, single site, brand-masked, non-dispensing, 2×2 bilateral crossover study. Each subject will be bilaterally fitted with one of the two test articles in each of the study periods.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Subjects between 18 and 39 (inclusive) years of age at the time of screening
  4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report.
  5. The subject must be willing to be photographed and/or video-taped.
  6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -5.00 D (inclusive) in each eye
  7. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye
  8. Have spherical best corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion).
  3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion).
  4. Any previous or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.).
  5. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment
  6. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician).
  7. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion).
  8. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VRC-East, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 subjects were enrolled into this study. Of those enrolled 25 were dispensed study lenses and completed the study, while 3 subjects failed to meet all eligibility criteria.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period.
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- All Subjects: All subjects who were dispensed a study lens.
Arm/Group | All Subjects
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (4.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Distance Binocular Visual Acuity (logMAR)
Description: Visual acuity on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters) under high luminance high contrast, high luminance low contrast and low luminance high contrast with distance goggles using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR value of 0.0 is equivalent to 20/20 Snellen vision.
Time Frame: 20- Minutes Post-Lens Fitting
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 25 | 25
logMAR
  High Luminance High Contrast | -0.15 (0.074) | -0.18 (0.069)
  High Luminance Low Contrast | 0.00 (0.083) | -0.04 (0.070)
  Low Luminance High Contrast with goggles | 0.02 (0.094) | 0.01 (0.065)

2. Primary Outcome: Near BinocularVisual Acuity (logMAR)
Description: Visual acuity on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at near (40 cm) under High luminance low contrast and low luminance high contrast with distance goggles using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR value of 0.0 is equivalent to 20/20 Snellen vision.
Time Frame: 20- Minutes Post-Lens Fitting
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Test | Control
Number analyzed (Participants) | 25 | 25
logMAR
  High Luminance Low Contrast | 0.04 (0.070) | 0.02 (0.076)
  Low Luminance High Contrast with goggles | -0.02 (0.072) | -0.04 (0.064)

3. Primary Outcome: Quantitative Visual Acuity
Description: Quantitative Visual Acuity (qVA) was measured at distance (4 meter) under low room illumination (4 lux), low luminance, high contrast conditions in the right eye only and in both eyes using AST Sentio vision Testing System. During testing 25 triplets of test letters were displayed on a large stationary monitor (118 CM), the operator recorded the patient's responses using the remote (Android Tablet). After a testing session had been completed the software calculated the VA threshold. VA threshold was defined as the logMAR stimulus size at which the expected probability of correct letter identification is 66%. when both eyes are measured. The average median VA threshold was reported for each lens. Lower values indicate better vision.
Time Frame: 20- Minutes Post-Lens Fitting
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 25 | 25
Number analyzed (eyes) | 50 | 50
logMAR
  Right Eye: number analyzed (eyes) | 25 | 25
  Right Eye | 0.061 (0.0889) | 0.051 (0.0749)
  Both Eyes | -0.010 (0.0578) | -0.039 (0.0645)

4. Primary Outcome: Area Under Contrast Sensitivity Function Curve
Description: Area under the log Curve was measured at 1.5, 3, 6, 12 and 18 cycles per degree (cpd) in the right eye only and in both eyes using AST Sentio vision Testing System. During testing 25 triplets of test letters were displayed on a large stationary monitor (118 CM), the operator recorded the patient's responses using the remote (Android Tablet). After a testing session had been completed the software calculated the Area under the log contrast sensitivity function from 1.5 cpd to 18 cpd. The average area under the log curve was reported for each lens. Higher values indicate better vision. Number of eyes is 50 when both eyes are measured.
Time Frame: 20- Minutes Post-Lens Fitting
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: log contrast sensitivity*cpd
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 25 | 25
Number analyzed (eyes) | 50 | 50
log contrast sensitivity*cpd
  Right Eye: number analyzed (eyes) | 25 | 25
  Right Eye | 1.254 (0.1746) | 1.273 (0.1584)
  Both Eyes | 1.524 (0.1092) | 1.535 (0.1022)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 day per subject.
Description: All subjects dispensed at least 1 study lens.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04287036/Prot_SAP_000.pdf